CLINICAL TRIAL: NCT06626828
Title: Acupuncture and Acupressure Treatment for Amnestic Mild Cognitive Impairment: a Pilot Randomized Controlled Trial
Brief Title: The Effect of Electroacupuncture Treatment on Cognitive Function in Adults With Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Prof Min Li, Dean and Chair Professor, School of Chinese Medicine, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/23-24/0234
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Amnestic Mild Cognitive Impairment - aMCI
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture group (Experimental): After sterilization, disposable sterilized needles (0.25 × 40 mm, Taichi disposable acupuncture needles, Suzhou Shenlong Medical Apparatus Company, Suzhou, China) are inserted by the Registered Chinese Medicine Practitioner (RCMP) into the acupoints of Shenting (GV24), left Benshen (GB13), right Benshen (GB13), Baihui (GV20), and Sishencong (EX-HN 1). Acupoints are then stimulated by the Huatuo SDZ-II electroacupuncture device.
  Interventions: Device: Electroacupuncture
- Control group (No Intervention): Blank control group with no further intervention.

INTERVENTIONS:
Device: Electroacupuncture — Disposable sterilized needles are inserted into selected acupoints at a depth of approximately 17-25 mm and an angle of 15-30° along the scalp. Acupoints are then stimulated by the SDZ-II electroacupuncture device, with a dilatational wave pattern at 4/20 Hz. The intensity of the stimulation was adjusted to the patient's tolerance.
  Arms: Electroacupuncture group

SUMMARY:
Background:

Amnestic mild cognitive impairment (aMCI) is a prevalent condition, often regarded as the transitional phase between normal cognitive aging and early Alzheimer's disease. Conventional treatments for aMCI remain limited, with pharmacological interventions showing mixed results and often failing to halt disease progression. Electroacupuncture (EA), is believed to improve cognitive function in various neurodegenerative disorders, including aMCI. Randomized controlled trials have also reported that acupuncture can positively influence cognitive function by promoting cerebral blood flow and modulating neurotransmitter activity, potentially offering a non-pharmacological approach to managing aMCI. However, robust clinical trials are lacking, and there is a need to assess the feasibility and efficacy of EA in treating aMCI. This pilot study aims to determine the preliminary efficacy of EA in improving cognitive function, and to evaluate the feasibility of the study design for future large-scale trials.

Methods:

This trial will be a multicenter, assessor- and data analyst-blind, pilot randomized controlled trial. A total of 24 participants aged 55-75 years, diagnosed with aMCI, will be recruited and randomly assigned in a 1:1 ratio into either the EA treatment group or a control group. Participants in the EA group will receive electroacupuncture at specific acupoints, while the control group will not undergo any intervention. The intervention will last 4 weeks, with two EA sessions per week, a total of 8 sessions. Assessments will be conducted at three time points: baseline, post-treatment (Week 4), and follow-up (Week 6). All participants will continue their standard medical care throughout the trial.

The primary outcome will be the change in cognitive function as measured by the Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA). Secondary outcomes will include changes in the Clinical Dementia Rating (CDR) and verbal fluency test, focusing on the memory domain. Safety and adverse events will be monitored throughout the study via follow-up assessments and questionnaires. Statistical analyses, including linear mixed models (LMM), will be performed using R and SPSS software, adhering to the intention-to-treat principle.

Expected Outcomes:

This pilot study is expected to provide preliminary data on the efficacy and safety of electroacupuncture in improving cognitive function in patients with aMCI. It will also assess the feasibility of conducting a larger-scale trial, including participant recruitment, adherence to the intervention, and the acceptability of outcome measures. Findings from this study will offer insights into the therapeutic potential of acupuncture and inform the design of future trials aimed at exploring its role as an alternative or complementary treatment for aMCI.

DETAILED DESCRIPTION:
Ethical Considerations:

Ethical approval for this study has been obtained from the Research Ethics Committee of Hong Kong Baptist University (REC/23-24/0234). All participants will provide written informed consent before enrollment, and their confidentiality and safety will be prioritized throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with an aMCI according to the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA)
2. With a Clinical Dementia Scale (CDR) score of 0.5, with the memory domain larger than 0
3. Within the age range of 55 to 75 years old
4. With visual and auditory acuity adequate for neuropsychological testing
5. Under a stable medical condition for 3 months prior to screening and baseline assessment
6. Under stable medications for 4 weeks before screening and baseline assessment

Exclusion Criteria:

1. With concurrent conditions that could contribute to the cognitive deficits, including any type of dementia including Alzheimer disease, vascular dementia, or any major psychiatric disorders such as major depressive disorder, schizophrenia, delirium, psychosis, etc.
2. With concurrent depression, anxiety, or suicidal thoughts within the past year
3. With concurrent major neurological conditions, including stroke, epilepsy and seizures, etc.
4. Currently immunocompromised due to receiving treatment for tumor, receiving immunosuppressive therapy, primary immunodeficiency, HIV infection, receiving high dose corticosteroids, etc
5. With bleeding disorders, including hemophilia, von Willebrand disease, vitamin K deficiency, etc.
6. With active neoplastic disease
7. Currently pregnant
8. Received acupuncture treatment for aMCI within a month before baseline assessment
9. Experienced severe allergy after receiving acupuncture treatment

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Domain and total score of the Hong Kong version of Montreal Cognitive Assessment (HK-MoCA) adjusted by age and education level | From baseline to Week 6
  Comprehensively evaluates multiple cognitive domains, including memory recall, visuospatial ability, language, attention, concentration, executive function, and orientation to time and space. The total score ranges from 0 to 30, with higher scores indicating better cognitive function. Scores are adjusted by age and education level. To mitigate the potential for practice effects, an alternate version of the HK-MoCA was employed during follow-up assessments.

SECONDARY OUTCOMES:
Clinical Dementia Rating (CDR) Sum of Boxes | From baseline to Week 6
  The CDR scale is a widely recognized and validated instrument used to assess the severity and stage of dementia by evaluating six key cognitive domains: memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care (Huang et al., 2021; O'Bryant et al., 2008). The overall CDR score ranges from 0 (normal cognition) to 3 (severe dementia), with higher scores indicating worse cognitive function. Specifically, a CDR-SoB score of 0.5-4.0 (corresponding to the overall CDR scores of 0.5), 4.5 to 9.0 (corresponding to the overall CDR scores of 1), 9.5 to 15.5 (corresponding to the overall CDR scores of 2), and 16.0 to 18.0 (corresponding to the overall CDR scores of 3) indicates MCI, mild, moderate, and severe dementia, respectively.
Verbal Fluency Test | From baseline to Week 6
  Verbal fluency was assessed by asking participants to recall as many words as possible within a specific semantic category in one minute, which serves as a measure of verbal executive function. For this study, animals and fruits were the categories used. The total number of words generated serves as the verbal fluency score, with higher scores indicating better verbal executive function. There is no predefined minimum or maximum for this test, but lower scores suggest impaired executive function and cognitive flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Baptist University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that support the findings in the publication, including demographics, patient characteristics, and outcome assessment data, etc. The anonymized datasets are available upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: From baseline to Week 6

REFERENCES:
- [Background] Tan TT, Wang D, Huang JK, Zhou XM, Yuan X, Liang JP, Yin L, Xie HL, Jia XY, Shi J, Wang F, Yang HB, Chen SJ. Modulatory effects of acupuncture on brain networks in mild cognitive impairment patients. Neural Regen Res. 2017 Feb;12(2):250-258. doi: 10.4103/1673-5374.200808. PMID 28400807
- [Background] Ma S, Huang H, Zhong Z, Zheng H, Li M, Yao L, Yu B, Wang H. Effect of acupuncture on brain regions modulation of mild cognitive impairment: A meta-analysis of functional magnetic resonance imaging studies. Front Aging Neurosci. 2022 Sep 23;14:914049. doi: 10.3389/fnagi.2022.914049. eCollection 2022. PMID 36212046
- [Background] He W, Li M, Han X, Zhang W. Acupuncture for Mild Cognitive Impairment and Dementia: An Overview of Systematic Reviews. Front Aging Neurosci. 2021 May 14;13:647629. doi: 10.3389/fnagi.2021.647629. eCollection 2021. PMID 34054504
- [Background] Yin Z, Li Y, Jiang C, Xia M, Chen Z, Zhang X, Zhao L, Liang F. Acupuncture for mild cognitive impairment: A systematic review with meta-analysis and trial sequential analysis. Front Neurol. 2023 Jan 6;13:1091125. doi: 10.3389/fneur.2022.1091125. eCollection 2022. PMID 36686535